CLINICAL TRIAL: NCT01867970
Title: RCT It's LiFe! to Evaluate the Effectiveness of the Monitoring and Feedback Tool and the Corresponding Counseling Protocol (Self-management Support Program) to be Executed by Practice Nurses in Primary Care
Brief Title: Interactive Tool to Support Self-management Through Lifestyle Feedback, Aimed at Physical Activity of COPD/DM Patients
Acronym: RCTIt'sLiFe!
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL42580.068.12; 40-00812-98-09025 (Other Grant/Funding Number: Zon Mw the Netherlands)
Record Dates: First submitted 2013-05-30; First posted 2013-06-04 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Chronic Obstructive Pulmonary Disease; Type 2 Diabetes
Keywords: remote sensing technology; physical activity; self-management support; primary care nursing
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Diabetes Mellitus, Type 2; Motor Activity | interventions — Equipment and Supplies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tool + Self-management Support Program (Experimental): The system consists of three elements: a 3D accelerometer worn on the hip together with; an application (app) on a smartphone; a server and a website. The patient receives three types of feedback on the mobile phone concerning the amount of activity, the amount of activity in relation to an activity goal, and the response of a nurse based on the measured activity. Practice nurses will use a consultation approach to coach patients in their self-management regarding physical activity based on a "five A's cycle" counselling technique (assess-advise-agree-assist-arrange). Motivational interviewing, risk assessment, and goal setting are specific aspects of this approach.The patient comes to the practice four times: in the first week, after 2 weeks, after 8-12 weeks and after 16-24 weeks.
  Interventions: Device: Tool; Behavioral: Self-management Support Program
- Self- management Support Program (Experimental): Practice nurses will use a consultation approach to coach patients in their self-management regarding physical activity based on a "five A's cycle" counselling technique (assess-advise-agree-assist-arrange). Motivational interviewing, risk assessment, and goal setting are specific aspects of this approach.The patient comes to the practice four times: in the first week, after 2 weeks, after 8-12 weeks and after 16-24 weeks.
  Interventions: Behavioral: Self-management Support Program
- Care as usual (No Intervention): Patients attend the practice regularly: at least once a year for a consultation with the GP. In addition, COPD patients have consultations (15-30 minutes) with the practice nurse once or twice a year. Most patients with diabetes type 2 see the GP ones per year and the practice nurse three times per year for a health check.Normally, physical activity is not high on the agenda during consultations with the practice nurse. Barriers for paying attention are the competition with other topics that should also be covered during consultations, co-morbidity and limitations of patients, and the assumption of most practice nurses that nowadays the patient decides on the topics of the consultation. All interviewees agreed that many patients do not perceive physical activity as an important issue.

INTERVENTIONS:
Device: Tool — The It's LiFe! tool consists of three different elements:
  1. the 3D accelerometer (Figure 7-8);
  2. the application (app) on a Samsung Smartphone (Figure 6);
  3. a web application and server called It's LiFe! online (powered by Sananet). The transmission of data from the accelerometer towards the app is via a Bluetooth connection. Every 15 minutes, or when the users press the refresh button, the Smartphone will connect to the accelerometer. The accelerometer should be within a 5 meter distance from the Smartphone. The transmission of data from the Smartphone towards the It's LiFe! server is via an internet connection. Therefore the Smartphone needs a SIM card with a data subscription.
  Other Names: MOX
  Arms: Tool + Self-management Support Program
Behavioral: Self-management Support Program — Consultations 1)The PN will increase awareness of the PA pattern, she will inform the patient about the health risks related to a sedentary lifestyle. Assessment of the PA level is done by completing the SQUASH questionnaire. The patient gets a leaflet with information about being active. 2)A day goal will be set in minutes a day, based on the results of the measurements of the first two weeks. The pre-measurement in condition 1 is an objective measurement by the tool and they are visible for the PN on the monitor portal of the It's LiFe! Server. The PN will encourage the patient to focus on goals that fit to the patient's preferences and to set up a SMART plan to reach personal goal. 3)The PN will discuss the results and barriers and facilitators related to physical activities. 4)The PN will discuss the results, behavior change and habits, with the patient.
  Arms: Self- management Support Program; Tool + Self-management Support Program

SUMMARY:
Rationale: Physical activity is an important factor for a healthy lifestyle. Although physical activity can delay complications and decrease the burden of the disease in chronically ill persons, their level of activity is often far from optimal. Many interventions have been developed to stimulate physical activity, with disappointing results. New in this field is the use of technology. Human persuasion (for example guidance by a practice nurse) can be enhanced by technological persuasion. Therefore a monitor and feedback tool, consisting of an accelerometer linked to a smart phone and webserver, has been developed and tested.

Objective: The main objective of this study is to measure the effects of the monitoring and feedback tool embedded in a Self-management Support Program on physical activity. The secondary objective is to measure the effect on self-efficacy, quality of life and health status. In addition a process evaluation will be conducted.

Study design: A three-armed cluster randomised controlled trial will be conducted with 240 patients from 24 general practices. Randomisation level is the practice. The following conditions will be compared: 1) Tool and Self-management Support Program; 2) Self-management Support Program; 3) Care as usual. Outcome measures will be measured at t0 (before the start of the intervention), t1 (after 6 months, at the end of the intervention) and t2 (after 9 months).

Study population: 120 People with COPD and 120 people with Diabetes type 2 (aged 40-70) treated in primary care will be included from 24 GP practices.

Intervention: Spread over a period of six months patients in condition 1 and 2 have to visit the practice nurse for 3-4 times for physical activity counselling. Specific activity goals will be set that are tailored to the individual patient's preferences and needs. On top of this, patients in condition 1 will be instructed to use the monitoring and feedback tool in daily life. Patients in condition 3 will not be exposed to any intervention.

Main study parameters/endpoints: Primary outcome: physical activity measured with a physical activity monitor (PAM). Secondary outcomes: quality of life, general self-efficacy, exercise self-efficacy and health status.

DETAILED DESCRIPTION:
A detailed study protocol is published Verwey, R., S. van der Weegen, et al. (2014). "A monitoring and feedback tool embedded in a counselling protocol to increase physical activity of patients with COPD or type 2 diabetes in primary care: study protocol of a three-arm cluster randomised controlled trial." BMC Family Practice 15(1): 93.

http://www.biomedcentral.com/1471-2296/15/93

ELIGIBILITY:
Inclusion Criteria:

* People diagnosed with COPD or diabetes type 2 who are predominantly treated in primary care and who benefit from more physical activity, will be included. -This means patients who do not comply with the Dutch Norm for Healthy Exercise (30 minutes activity per day of a moderate intensity during five days a week)
* Their age should be between 40-70 years to ensure homogeneity in the groups
* Additional inclusion criteria for the diabetes group are a recent (no longer than a year ago) HbA1c concentration of more than 7% / more than 53 mmol/mol and a body mass index of more than 25kg/m2

For the COPD group the following additional inclusion criteria apply:

-A clinical diagnosis of COPD according to the GOLD-criteria stage 1, 2 and 3 (post bronchodilator FEV1/IVC <= 70% and FEV1 between 30 and 80% of the predicted value); at least six weeks respiratory stable and on a stable drug regimen

Exclusion Criteria:

-Patients older than 70 years are not included because of a bigger risk for co-morbidity and a higher chance of mobility problems (balance)

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2013-04; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Physical activity | Change between baseline (T0) and directly after the intervention, after 4-6 months from baseline (T1)
  Physical activity will be measured with the Personal Activity Monitor (PAM). The PAM is a small (58 x 42 x 13 mm, weight 28 gram) tri-axial accelerometer that can be easily attached to a belt and is worn on the hip. The PAM registers all movements that are made on a day and measures the intensity of hip movements. Via a docking station, which must be connected to the internet, the PAM scores can be uploaded and converted into minutes a day in a sedentary category (< 1.8 METS) a living category (1.8-3 METS) a moderate category (3-7 METS) and a vigorous category (>7 METS). The number of minutes of physical activity in the moderate and vigorous category is used as an outcome measurement. The possibility of noticing (e.g. providing feedback) users about their activity scores and their calories used will be deactivated; the displays will be turned off. The level of physical activity in minutes a day at t0 will be compared to the minutes of activity at t1 and t2.
Physical activity | Change between T1 and T2: 3 months follow up
  Physical activity will be measured with the Personal Activity Monitor (PAM). The PAM is a small (58 x 42 x 13 mm, weight 28 gram) tri-axial accelerometer that can be easily attached to a belt and is worn on the hip. The PAM registers all movements that are made on a day and measures the intensity of hip movements. Via a docking station, which must be connected to the internet, the PAM scores can be uploaded and converted into minutes a day in a sedentary category (< 1.8 METS) a living category (1.8-3 METS) a moderate category (3-7 METS) and a vigorous category (>7 METS). The number of minutes of physical activity in the moderate and vigorous category is used as an outcome measurement. The possibility of noticing (e.g. providing feedback) users about their activity scores and their calories used will be deactivated; the displays will be turned off. The level of physical activity in minutes a day at t0 will be compared to the minutes of activity at t1 and t2.

SECONDARY OUTCOMES:
Quality of life | Change between baseline (T0) and directly after the intervention, after 4-6 months from baseline (T1)
  To measure the quality of life of participants the Dutch version of the SF-36 will be used (see appendix F1.3). The SF-36 is a generic health status instrument designed for the use across a wide range of chronic disease populations. "The SF-36 has shown an excellent reliability and validity in diverse patient populations in the US and the Netherlands. The SF-36 is composed of 36 items, organized into 8 multi-item scales covering a similar number of dimensions, including physical functioning, physical role functioning, bodily pain, general health, vitality, social functioning, emotional role functioning, and mental health.". A higher score on the SF-36 indicates a better quality of life.
(General and Exercise) Self-efficacy | Change between baseline (T0) and directly after the intervention, after 4-6 months from baseline (T1)
  Self-efficacy is described as people's belief in their capability to organize and execute the course of action required to deal with prospective situations. Self-efficacy is an important construct since it influences the processes of planning, taking initiative, maintaining behaviour change, and managing relapses.
  To measure self-efficacy of participants two questionnaires will be used: the Dutch adaptation of the General Self-Efficacy Scale (GSE) from Jerusalem and Schwarzer (1995) and the Dutch adaptation of the Exercise Self-efficacy Scale (ESS) developed by Bandura (1997). The GSE contains 10 questions in a 4 points response format and the ESS contains 18 questions regarding different situations related to exercise with a scale response format from 0-100.
Health status | Change between baseline (T0) and directly after the intervention, after 4-6 months from baseline (T1)
  Personal reported health status will be measured by a disease specific questionnaire.
  For diabetes the Diabetes Symptom Checklist-revised (DSC-R) will be used. On the 34 items of the DSC-R, participants first indicate whether they have experienced each symptom in the past 4 weeks. If "yes" is selected, the participant continues to rate how troublesome that symptom is on a 5-point scale ranging from 1 (not at all) to 5 (extremely). The instrument yields a total score and the following subscales: Fatigue, Cognitive, Pain, Sensory, Cardiology, Ophthalmology, Hypoglycemia, and Hyperglycemia. The total score and all dimension scores range from 0 to 5. Higher scores indicate greater symptom burden.
  For COPD the Chronic Respiratory Questionnaire (CRQ) will be used. The CRQ consists of four domains: fatigue, dyspnoea, mastery (the patient's feeling of control over their disease), and emotional function.
Quality of life | Change between T1 and T2: 3 months follow up
  To measure the quality of life of participants the Dutch version of the SF-36 will be used (see appendix F1.3). The SF-36 is a generic health status instrument designed for the use across a wide range of chronic disease populations. "The SF-36 has shown an excellent reliability and validity in diverse patient populations in the US and the Netherlands. The SF-36 is composed of 36 items, organized into 8 multi-item scales covering a similar number of dimensions, including physical functioning, physical role functioning, bodily pain, general health, vitality, social functioning, emotional role functioning, and mental health.". A higher score on the SF-36 indicates a better quality of life.
(General and Exercise) Self-efficacy | Change between T1 and T2: 3 months follow up
  Self-efficacy is described as people's belief in their capability to organize and execute the course of action required to deal with prospective situations. Self-efficacy is an important construct since it influences the processes of planning, taking initiative, maintaining behaviour change, and managing relapses.
  To measure self-efficacy of participants two questionnaires will be used: the Dutch adaptation of the General Self-Efficacy Scale (GSE) from Jerusalem and Schwarzer (1995) and the Dutch adaptation of the Exercise Self-efficacy Scale (ESS) developed by Bandura (1997). The GSE contains 10 questions in a 4 points response format and the ESS contains 18 questions regarding different situations related to exercise with a scale response format from 0-100.
Health status | Change between T1 and T2: 3 months follow up
  Personal reported health status will be measured by a disease specific questionnaire.
  For diabetes the Diabetes Symptom Checklist-revised (DSC-R) will be used. On the 34 items of the DSC-R, participants first indicate whether they have experienced each symptom in the past 4 weeks. If "yes" is selected, the participant continues to rate how troublesome that symptom is on a 5-point scale ranging from 1 (not at all) to 5 (extremely). The instrument yields a total score and the following subscales: Fatigue, Cognitive, Pain, Sensory, Cardiology, Ophthalmology, Hypoglycemia, and Hyperglycemia. The total score and all dimension scores range from 0 to 5. Higher scores indicate greater symptom burden.
  For COPD the Chronic Respiratory Questionnaire (CRQ) will be used. The CRQ consists of four domains: fatigue, dyspnoea, mastery (the patient's feeling of control over their disease), and emotional function.
Physical activity in daily life | Change between baseline (T0) and directly after the intervention, after 4-6 months from baseline (T1)
  The PAM scores and the number of minutes of PA in the living, moderate and vigorous category >1.8 METS. These measures indicate all types of activity during the day.
Physical activity in daily life | Change between T1 and T2: 3 months follow up
  The PAM scores and the number of minutes of PA in the living, moderate and vigorous category >1.8 METS. These measures indicate all types of activity during the day.

OTHER OUTCOMES:
Health status | Change between baseline (T0) and directly after the intervention, after 4-6 months from baseline (T1)
  If available in the medical record of the general practitioner, disease specific health outcomes will be extracted, such as CCQ, MRC values for COPD patients and Hba1C blood values for diabetes patients, blood pressure and BMI.
Health status | Change between T1 and T2: 3 months follow up
  If available in the medical record of the general practitioner, disease specific health outcomes will be extracted, such as CCQ, MRC values for COPD patients and Hba1C blood values for diabetes patients, blood pressure and BMI.

CONTACTS AND LOCATIONS:
Locations (1):
- Luc de Witte, Maastricht, Netherlands

REFERENCES:
- [Derived] van der Weegen S, Verwey R, Spreeuwenberg M, Tange H, van der Weijden T, de Witte L. It's LiFe! Mobile and Web-Based Monitoring and Feedback Tool Embedded in Primary Care Increases Physical Activity: A Cluster Randomized Controlled Trial. J Med Internet Res. 2015 Jul 24;17(7):e184. doi: 10.2196/jmir.4579. PMID 26209025
- [Derived] Verwey R, van der Weegen S, Spreeuwenberg M, Tange H, van der Weijden T, de Witte L. A monitoring and feedback tool embedded in a counselling protocol to increase physical activity of patients with COPD or type 2 diabetes in primary care: study protocol of a three-arm cluster randomised controlled trial. BMC Fam Pract. 2014 May 12;15:93. doi: 10.1186/1471-2296-15-93. PMID 24885096